CLINICAL TRIAL: NCT03786965
Title: Evaluating of Role of Myeloperoxidase in Prediction of Outcomes of Cardiac Surgery Procedures.
Acronym: MPO-CSP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Aleksandr Nemkov, PhD, St. Petersburg State Pavlov Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: №22/18-H
Record Dates: First submitted 2018-12-20; First posted 2018-12-26 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-11

CONDITIONS: Cardiac Procedure Complication; Ischemic Heart Disease; Valve Heart Disease; Defect Septal
Keywords: Ischemic Heart Disease; Valve Disease; Septal Defect; Myeloperoxidase; Molecular biology; Gene analysis
MeSH Terms: conditions — Myocardial Ischemia; Heart Valve Diseases; Heart Septal Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- On-pump CABG. (Other): On-pump CABG.
  Interventions: Other: On-pump CABG
- Off-pump CABG. (Other): Off-pump CABG.
  Interventions: Other: Off-pump CABG
- Pump-assisted CABG. (Other): Pump-assisted CABG.
  Interventions: Other: Pump-assisted CABG
- Heart Valve Procedure without CABG. (Other): Heart Valve Procedure without CABG.
  Interventions: Other: Valve Repair Procedure without CABG.
- Heart Valve Procedure with CABG. (Other): Heart Valve Procedure with CABG.
  Interventions: Other: Valve Repair Procedure with CABG.

INTERVENTIONS:
Other: On-pump CABG — On-pump CABG
  Arms: On-pump CABG.
Other: Off-pump CABG — Off-pump CABG
  Arms: Off-pump CABG.
Other: Pump-assisted CABG — Pump-assisted CABG
  Arms: Pump-assisted CABG.
Other: Valve Repair Procedure without CABG. — Valve Repair Procedure without CABG (open heart procedure).
  Arms: Heart Valve Procedure without CABG.
Other: Valve Repair Procedure with CABG. — Valve Repair Procedure with CABG (open heart procedure).
  Arms: Heart Valve Procedure with CABG.

SUMMARY:
The main objection is to investigate molecular biology of myocardial damage during cardiac surgery procedures.

DETAILED DESCRIPTION:
To assess outcomes after cardiac surgery procedures. To investigate serum level of myeloperoxidase, morphology of left atrium appendage, to perform genetic analysis and cell biology.

ELIGIBILITY:
Inclusion Criteria:

* ischemic heart disease with indications for operation
* valve disease with indications for operation
* ischemic heart disease combined with valve disease with indications for operation

Exclusion Criteria:

* patient refusal

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2025-07-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Death within 30 days after procedure. | within 30 days after procedure.
  Death within 30 days after surgical procedure.
Acute myocardial infarction. | within 30 days after procedure.
  Acute myocardial infarction (ST-changes with troponin I > 10 ng/ml).
Stroke. | within 30 days after procedure.
  Stroke (MRI changes or corresponding neurologist record).
Arrhythmia | within 30 days after procedure.
  Any type of arrhythmia including AV-block.
Renal dysfunction. | within 30 days after procedure.
  Renal dysfunction if serum creatinine greater than 25% of upper reference range.
Infection or febrile. | within 30 days after procedure.
  Infection or febrile (t> 37 or CRP elevation or long regeneration of surgical wound).
Respiratory dysfunction. | within 30 days after procedure.
  Respiratory dysfunction (pulmonary ventilation longer than 2 days).

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Nemkov, PhD, Study Director — First Saint-Petersburg Medical University
Locations (1):
- Nikolai Bunenkov, Saint Petersburg, Non-US/Non-Canadian, Russia

IPD SHARING:
Plan to Share IPD: No
Individual participant data are confidential.